CLINICAL TRIAL: NCT06269133
Title: Evaluating the Safety and Effectiveness of Cemiplimab in Combination With Platinum-Doublet Chemotherapy by Demographic Characteristics in First-Line Treatment of Advanced Non-Small Cell Lung Cancer: A Multi-Database Real World Evidence Study in US Patients
Brief Title: Evaluation of Cemiplimab in Combination With Platinum-Doublet Chemotherapy in First-Line (1L) Treatment of Advanced Non-Small Cell Lung Cancer (NSCLC) in Adult United States (US) Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R2810-ONC-22115
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Advanced Non-small Cell Lung Cancer
Keywords: Advanced non-small cell lung cancer (aNSCLC); Epidermal growth factor receptor (EGFR); Anaplastic lymphoma kinase (ALK); C-ros oncogene receptor tyrosine kinase (ROS1)
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Patients: Patients who have received cemiplimab in combination with platinum-doublet chemotherapy for the 1L treatment of aNSCLC in the US with no documented EGFR, ALK and ROS1 variants as described in the protocol.
  Interventions: Drug: REGN2810; Other: Platinum-doublet chemotherapy

INTERVENTIONS:
Drug: REGN2810 — No study specific interventions for this non-interventional-observational study; patients had previously been administered this treatment.
  Other Names: LIBTAYO®; cemiplimab
Other: Platinum-doublet chemotherapy — No study specific interventions for this non-interventional-observational study; patients had previously been administered this treatment.

SUMMARY:
This multi-year cohort study will assess the real-world safety and effectiveness of 1L treatment with cemiplimab in combination with platinum-doublet chemotherapy across advanced NSCLC patient subgroups defined by age, sex, race, and ethnicity. Patients will be retrospectively identified from at least two US electronic health record (EHR)-based databases.

DETAILED DESCRIPTION:
Patients and baseline variables will be captured retrospectively, but outcome measures will be prospectively ascertained.

ELIGIBILITY:
Key Inclusion Criteria:

1. Advanced non-small cell lung cancer (aNSCLC) (defined as stage IIIB/C or stage IV) treated with cemiplimab in combination with platinum-doublet chemotherapy in the 1L setting from Nov 2022 to Jun 2026 as described in the protocol

Key Exclusion Criteria:

1. Patients who have EGFR, ALK or ROS1 variants
2. Treatment with EGFR, ALK or ROS1 inhibitors at any time prior to the index date
3. Patients actively enrolled in a clinical trial in which they receive treatment with cemiplimab in combination with platinum-doublet chemotherapy

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced disease, defined as stage IIIB, IIIC, or IV disease, with evidence of administration of 1L cemiplimab in combination with platinum-doublet chemotherapy between 08 Nov 2022 and 30 Jun 2026 and without EGFR, ALK, or ROS1 genomic variants, or actively enrolled in a clinical trial in which they receive treatment with cemiplimab in combination with platinum-doublet chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-23 (Estimated)

PRIMARY OUTCOMES:
Real-world response rate (rwRR) | Approximately 3 years
Any treatment-emergent immune-mediated adverse event (imAE) | Approximately 3 years
Any treatment-emergent imAE resulting in hospitalization | Approximately 3 years
Any treatment-emergent imAE resulting in death | Approximately 3 years
Specific treatment-emergent imAEs | Approximately 3 years

SECONDARY OUTCOMES:
Real-world duration of response (rwDOR) | Approximately 3 years
Real-world progression-free survival (rwPFS) | Approximately 3 years
Real-world overall survival (rwOS) | Approximately 3 years
Treatment-emergent immune-mediated adverse events (imAEs) | Approximately 3 years
Infusion-related reaction (IRR) | Approximately 3 years
IRR resulting in hospitalization | Approximately 3 years
IRR resulting in death | Approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Research Facility, Tarrytown, New York, United States